CLINICAL TRIAL: NCT05696470
Title: Fusion Rates of 3D Printed Porous Titanium Cages in Three and Four Level ACDFs
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Andrew Grossbach, Assistant Clinical Professor Residency Program Director Deformity and Robotic Spinal Fellowship Director, Ohio State University
Other Study IDs: 2020H0309
Record Dates: First submitted 2022-10-18; First posted 2023-01-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Radiculopathy; Myelopathy Cervical; Foraminal Stenosis; Central Canal Stenosis
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: DePuy Synthes Conduit 3D printed titanium cages — DePuy Conduit 3D printed titanium cages supplemented with SKYLINE Anterior Cervical Plate System and 1 CC DBM

SUMMARY:
The purpose of this trial is to assess fusion rates in 3 and 4 level ACDFs in patients implanted with DePuy Conduit 3D printed titanium cages supplemented with SKYLINE Anterior Cervical Plate System and 1 CC DBM. This will be a non-inferiority study, looking to show that Synthes Conduit 3D printed titanium cages fuse as well as cages.

DETAILED DESCRIPTION:
This is a prospective, single arm study of clinical and radiological outcomes from anterior cervical discectomy and fusions for cervical spondylosis. 58 Patients undergoing 3 to 4 level ACDF procedures from C2-T1 will be enrolled. Patients will be implanted with DePuy Conduit Titanium ACDF cage (DePuy Synthes, Raynham, MA). A retrospective comparision group will be used. The retrospective group will include 58 consecutive patients undergoing 3-4 level ACDFs with milled allograft.

This single-centered study will enroll up to 58 subjects, with subjects followed for 24 months post-surgery. All subjects enrolled in the study will be recruited from a pool of subjects eligible for three or four level anterior cervical fusion surgeries. The inclusion/exclusion criteria are listed below.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Symptomatic multi-level degenerative cervical spondylosis necessitating anterior cervical arthrodesis in the subaxial cervical spine (between C2-T1).
* Surgery performed within the Department of Neurological Surgery at The Ohio State University Wexner Medical Center (OSUWMC)
* Cervical x-rays at 24 months (±60 days; retrospective comparison group only)

Exclusion Criteria:

* Traumatic spinal fractures or spinal cord injury
* Previous cervical fusion surgery
* Co-morbidity requiring medication use that may interfere with bone or soft tissue healing (i.e., high dose oral or parenteral glucocorticoids, immunosuppressive agents, methotrexate) - at discretion of investigator
* Severe co-morbidities (e.g., heart, respiratory, or renal disease)
* Recent (<3 yrs) or co-incident spinal tumor or infection
* Concurrent involvement in another investigational drug or device study that could confound study data (prospective exclusion only)
* History of substance abuse (recreational drugs, prescription drugs or alcohol) that could interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up
* Subjects who are pregnant or plan to become pregnant in the next 24 months
* Prisoner
* Other contraindications for DePuy Conduit 3D printed titanium cage implant (prospective exclusion only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing 3 to 4 level ACDF procedures from C2-T1
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fusion rate | 24 months
  based on postoperative X-ray: presence of bone trabeculae across graft-host interface, absence of radiolucent gap between graft and adjacent vertebral body, restriction of motion to 2mm or less between adjacent vertebral spinous processes on flexion-extension lateral radiographs

SECONDARY OUTCOMES:
NRS | 24 months
  Numeric Rating Scale for neck and arm pain
NDI | 24 months
  Neck Disability Index
SF36 RAND | 24 months
  Short Form 36 RAND
Neurological assessment: Upper Extremity Strength | 24 months
  grip, biceps, triceps, delts, intrinsics, wrist extrinsic) measured on scale of 0-5 follwing INSCI assessment for Manual Muscle Testing (MMT)
Cervical sagittal alignment | 24 months
  Standing radiographs of the sagittal spine to identify changes in functional sagittal; will measure the Cobb angle between the lower endplate of C2 and C7 (C2L-C7L angle) alignment after cervical fusion as determined by functional segments between cervicothoracic and thoracolumbar. Patient cervical 4 view x-rays pre-operatively and at follow-ups will be compared.
Reoperation | 24 months
  Reoperation at cervical and thoracic levels while patient is enrolled in the study. Hardware removed, new hardware added
number of days in the hospital | up to 24 months
  number of days in the hospital
Adverse events | 24 months
  wound infection, dysphagia, hematoma, dysphonia, DVT, etc
Neurological assessment: Sensory function (C2-C7 dermatome) | 24 months
  Pin prick sensation is assessed with a needle. Light touch sensation is assessed with a piece of tissue paper.
Neurological assessment: Sensation is scored as absent (0), abnormal (1), or normal (2) | 24 months
  Reflexes (Biceps, Brachioradials, Triceps)-Upper and lower extremities should be examined for asymmetry in deep tendon reflexes.
Neurological assessment: Hoffman's and Spurlings | 24 months
  Testing for positive or negative indication

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center Neurological Surgery, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided